CLINICAL TRIAL: NCT04714658
Title: Efficiency of a Therapeutic Patient Education Program in Myasthenia Gravis
Brief Title: Education Program in Myasthenia
Acronym: MG-ETP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7534
Record Dates: First submitted 2020-11-25; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-11

CONDITIONS: Auto-immune Myasthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate PTE (Experimental)
  Interventions: Other: Therapeutic Education
- 6-month deferred PTE (Other)
  Interventions: Other: Therapeutic Education

INTERVENTIONS:
Other: Therapeutic Education — Each patient will participate in 1 to 3 PTE sessions.
  1. st group collective workshop : allow the patient to better understand autoimmune
  2. nd workshop : fatigue and techniques that enable its best management.
  3. rd workshop : improving the management of the emotions generated by myasthenia. It allows patients to express their experiences of the disease in front of a group, to talk about their difficulties in their relationships and mobilize their resources to promote exchanges.

SUMMARY:
Patient therapeutic education (PTE) has become "a must" in the modern management of chronic diseases. Its main objective is to improve compliance with treatment and the application of preventive measures. The main goal of this study is to assess the influence of the therapeutic education program on the perception of the disease in patients with autoimmune myasthenia. Secondary objectives are to assess quality of life, patient satisfaction of the PTE program, the acquisition of therapeutic goals and the influence of therapeutic education on the evolution of autoimmune myasthenia Study team hypothesize that therapeutic education could improve the patient's perception of myasthenia and its quality of life. By improving patient's adherence to treatments and his knowledge of the disease, it could also improve the evolution of myasthenia gravis. Study team suppose that PTE program can reduce the absenteeism at work, the number and duration of hospitalizations, particularly those in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Patient with generalized autoimmune myasthenia with Acetylcholine Receptor Antibodies (AChR Ab) or with antibodies to the muscle-specific receptor tyrosine kinase (MuSK Ab)
* Patient agreeing to participate in the therapeutic education program
* Signing consent
* Subject affiliated with a health insurance social protection regiment

Exclusion Criteria:

* Patients without serological confirmation of myasthenia or pure ocular form
* Patient with cognitive impairment or behavioral problems that, in the investigator's opinion, will compromise their ability to comply with study procedures
* Refusal of the patient to participate in the study
* Patient who has already benefited from the therapeutic education program in myasthenia
* Age < 18 y.o.
* Subject under safeguarding justice
* Subject under guardianship or under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-22 (Estimated); Primary Completion 2025-05-22 (Estimated); Study Completion 2025-05-22 (Estimated)

PRIMARY OUTCOMES:
Brief Illness Perception Questionnaire | 6 month after the first visit

IPD SHARING:
Plan to Share IPD: No